CLINICAL TRIAL: NCT04896437
Title: Direct Use of Autologous Fat Graft on The Treatment of Lower Extremity Wounds
Brief Title: Direct Use of Non-centrifuged Autologous Fat Graft
Status: Completed | Type: Observational
Sponsor: Samsun Liv Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Retrospective study
Record Dates: First submitted 2021-05-06; First posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Wound Healing Delayed
Keywords: diabetic food; lower extremity; fat graft; nonentrifuged

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: non-centrifuge fat graft application to the wounds — Autologous fat grafts were harvested from abdominal or gluteal regions of the patients and injected into the wound bed and wound environment. Clinical observation and photograph records were used to follow the wounds.

SUMMARY:
There are a limited number of reports related to the direct use of non-centrifuged adipose tissue graft in the literature. This preliminary study aims to present our experience on the efficacy of autologous fat graft use without centrifuging in the treatment of lower extremity wounds.

DETAILED DESCRIPTION:
16 wounds treated with non-centrifuged autologous fat grafts were included in the study. The data were retrospectively analyzed. VAC (vacuum-assisted therapy) or silver-impregnated dressing was used to achieve a healthy wound bed before fat grafting. Autologous fat grafts were harvested from abdominal or gluteal regions of the patients and injected into the wound bed and wound environment. Clinical observation and photograph records were used to follow the wounds.

ELIGIBILITY:
Inclusion Criteria:

1. diabetic,
2. venous
3. traumatic wounds

Exclusion Criteria:

1. Malignancy,
2. A life expectation <1 year,
3. Chemical or radiation exposure.
4. Pregnancy

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 16 lower extremity wounds were included in the study between January 2016-October 2019 years. All patients were treated by two surgeons in the same clinic. The wounds were those that continued for at least three months of high to moderate exudate and required open management of the secondary intervention. The etiologies of the wounds were diabetic, venous or traumatic ulcers.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
Wounds examination | 6 months
  Collection of the data from clinical observation and photograph records were made to follow the wounds. the observations were made during changing the wound dressing and generally every three days.

SECONDARY OUTCOMES:
Wounds classification according to data from files and photographs | 3 months
  In this season the data will be classified according to the wounds parameters and photograph
Final evaluation and data achieving from files and exam carts | 3 months
  all data will be examined and evaluated whether there is any difference between probable groups

CONTACTS AND LOCATIONS:
Overall Officials: Umut Tuncel, Assoc Prof, Principal Investigator — Samsun Liv Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goncalves AI, Gershovich PM, Rodrigues MT, Reis RL, Gomes ME. Human adipose tissue-derived tenomodulin positive subpopulation of stem cells: A promising source of tendon progenitor cells. J Tissue Eng Regen Med. 2018 Mar;12(3):762-774. doi: 10.1002/term.2495. Epub 2017 Oct 4. PMID 28593712
- [Background] Hivernaud V, Lefourn B, Robard M, Guicheux J, Weiss P. Autologous fat grafting: A comparative study of four current commercial protocols. J Plast Reconstr Aesthet Surg. 2017 Feb;70(2):248-256. doi: 10.1016/j.bjps.2016.11.022. Epub 2016 Dec 14. PMID 28043786
- [Background] Conde-Green A, Marano AA, Lee ES, Reisler T, Price LA, Milner SM, Granick MS. Fat Grafting and Adipose-Derived Regenerative Cells in Burn Wound Healing and Scarring: A Systematic Review of the Literature. Plast Reconstr Surg. 2016 Jan;137(1):302-312. doi: 10.1097/PRS.0000000000001918. PMID 26710034
- [Background] Tuncel U, Kostakoglu N, Turan A, Cevik B, Cayli S, Demir O, Elmas C. The Effect of Autologous Fat Graft with Different Surgical Repair Methods on Nerve Regeneration in a Rat Sciatic Nerve Defect Model. Plast Reconstr Surg. 2015 Dec;136(6):1181-1191. doi: 10.1097/PRS.0000000000001822. PMID 26273733
- [Background] Moyer HR, Namnoum JD. Autologous Fat Transfer: The Progenitor Cell Response to Different Recipient Environments. Aesthet Surg J. 2014 Aug;34(6):932-40. doi: 10.1177/1090820X14536903. Epub 2014 Aug 1. PMID 24936093
- [Background] Hyldig K, Riis S, Pennisi CP, Zachar V, Fink T. Implications of Extracellular Matrix Production by Adipose Tissue-Derived Stem Cells for Development of Wound Healing Therapies. Int J Mol Sci. 2017 May 31;18(6):1167. doi: 10.3390/ijms18061167. PMID 28561757
- [Background] van de Vyver M. Intrinsic Mesenchymal Stem Cell Dysfunction in Diabetes Mellitus: Implications for Autologous Cell Therapy. Stem Cells Dev. 2017 Jul 15;26(14):1042-1053. doi: 10.1089/scd.2017.0025. Epub 2017 May 18. PMID 28447876
- [Background] Hur W, Lee HY, Min HS, Wufuer M, Lee CW, Hur JA, Kim SH, Kim BK, Choi TH. Regeneration of full-thickness skin defects by differentiated adipose-derived stem cells into fibroblast-like cells by fibroblast-conditioned medium. Stem Cell Res Ther. 2017 Apr 20;8(1):92. doi: 10.1186/s13287-017-0520-7. PMID 28427476